CLINICAL TRIAL: NCT04389528
Title: Evaluation of the Effect of tDCS on Cannabis Craving: Multicentre Randomized, Double-blind Study Versus Placebo
Brief Title: Evaluation of the Effect of tDCS on Cannabis Craving
Acronym: TCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Januel (Other)
Responsible Party: Sponsor-Investigator, Januel, Head of the clinical research unit of ville evrard, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 10477M-TCC
Record Dates: First submitted 2020-04-27; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Addiction to Cannabis

STUDY DESIGN:
Intervention Model Description: double-blind randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS active arm (Experimental)
  Interventions: Other: Neuromodulation by tDCS
- tDCS placebo (Placebo Comparator)
  Interventions: Other: Neuromodulation by tDCS

INTERVENTIONS:
Other: Neuromodulation by tDCS — The tDCS is a device for modulating cortical excitability. It consists of passing a low intensity direct electrical current over the scalp via two electrodes: an anode and a cathode soaked in a saline solution. Although there is a short-circuit effect through the scalp, a significant amount of electrical current enters the brain and changes the transmembrane potential.

SUMMARY:
Cannabis is the most frequently consumed drug in France and its use continues to increase. Over the 18-64 age group as a whole, experimentation with cannabis at least once in a lifetime increased from 33% in 2010 to 42% in 2014, confirming the upward trend observed since the 1990.

Cannabis, like all drugs, disrupts the reward circuit whose neurons originate in the ventral tegmental area and project into the mesolimbic and cortical structures.

Acute cannabis use is thought to increase mesolimbic dopamine by affecting the Gabaergic or Glutamatergic system.

Chronic cannabis use usurps the reward system and leads to changes in the mesolimbic circuit (nucleus accumbens, ventral tegmental area, amygdala, and prefrontal cortex), inducing increased craving, with persistent craving for the substance and vulnerability to relapse.

Cognitively, addiction is associated with increased impulsivity, with a propensity to take risks leading to impaired decision-making.

There is currently no validated drug treatment for cannabis addiction. Non-invasive brain stimulation could be an interesting therapeutic alternative.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between 18 and 65 years of age
2. Right-Handers
3. Diagnosis: Cannabis Use Disorder (according to DSM 5 criteria)
4. Patient with no other drug or psychotherapeutic treatment for cannabis addiction ("naive" patients)
5. Reported use of cannabis more than three times a week in the past three years
6. Signing consent to participate in research

Exclusion Criteria:

1. Pregnancy or lack of effective contraception
2. Patients with severe somatic disease
3. Other addictions of "moderate" to "severe" intensity according to DSM 5 criteria (excluding tobacco and coffee)
4. Patients undergoing antidepressant or neuroleptic or thyroid-regulating therapy.
5. Contraindications to tDCS (presence of an intracranial metal body, intracranial hypertension)
6. Topic that has already been stimulated by tDCS
7. Patients under reinforced guardianship or curatorship

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-07-17 (Estimated); Study Completion 2021-12-17 (Estimated)

PRIMARY OUTCOMES:
Evaluating the change from craving to cannabis. by an analog visual scale .Scores (0 to 10) | 3 months

SECONDARY OUTCOMES:
The change to cannabis craving assessed by the Baseline Marijuana Craving Test at the end of treatment | 3 month
The change in cannabis craving during an incentive to use task evaluated by analog visual scale scores (0 to 10) | 3 months
Montgomery-Åsberg depression rating scale) Scores (0 to 60) | 3 months
evaluation of the change in the number of joints consumed per day | 3 months
evaluation of the change in the number of cigarettes consumed per day | 3 months
assessment of the change in attention and inhibition skills as assessed by the Stroop test before and after a neurofeedback test | 3 months
the Gambling Task's assessment of decreased risk-taking | 3 months
Young Mania Rating Scale Scores (0 to 60) | 3 months
Beck Depression Inventory Scores (0 to 39) | 3 months
Clinical Global Impression Severity of disease (0 to 7) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Noomane BOUAZIZ, Principal Investigator — Clinical Unite research of EPS Ville Evrard
Locations (1):
- Youcef BENCHERIF, Maisons-Alfort, Île-de-France Region, France